CLINICAL TRIAL: NCT06980311
Title: Comparison of the Effects of Music Therapy-Based Aerobic Exercise and Traditional Aerobic Exercise Training on Cardiopulmonary Functions, Functional Capacity, Balance, Peripheral Muscle Strength, Cognitive Functions, Depression, and Quality of Life in Geriatrics
Brief Title: Comparing Music-Supported and Traditional Aerobic Training in Geriatric Health Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Gökhan Can TÖRPÜ, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02.05.2025-BezmialemVU
Record Dates: First submitted 2025-05-02; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Geriatric; Aerobic Exercise; Music Therapy; Physiotherapy and Rehabilitation
MeSH Terms: interventions — Exercise; Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Aerobic Exercise Training Group (Active Comparator): Traditional Aerobic Exercise group will undergo treadmill-based aerobic exercise training under the supervision of a physiotherapist twice a week for a total of 8 weeks.
  Interventions: Other: Aerobic Exercise
- Music Therapy-Based Aerobic Exercise Training Group (Experimental): Music Therapy-Based Aerobic Exercise Training group will follow the same treadmill exercise program as the Traditional Aerobic Exercise group. However, during the exercise sessions, music therapy will be applied according to the beats per minute (BPM) ranges.
  Music will be used throughout the exercise sessions to regulate participants' heart rate and blood pressure, reduce perceived fatigue, enhance motivation, and support rhythmic movement patterns. During training, participants' heart rate and oxygen saturation will be monitored using a fingertip pulse oximeter.
  Interventions: Other: Aerobic exercise with music therapy
- Control Group (No Intervention): Individuals in the control group will be provided with physical activity counseling in line with the physical activity guidelines recommended by the World Health Organization (WHO). Participants will be advised to do at least 150-300 minutes of moderate-intensity aerobic physical activity per week and will be informed about the positive effects of movement on health. Participants will continue their current medical treatments (if any) in accordance with the recommendations of their physicians. All participants will be evaluated at the beginning and end of the study.

INTERVENTIONS:
Other: Aerobic Exercise — Traditional Aerobic Exercise group will undergo treadmill-based aerobic exercise training under the supervision of a physiotherapist twice a week for a total of 8 weeks. For participant safety, they will be instructed to hold onto the handrails while walking, and proper use of the safety key will be ensured during each session.
  Using the ULTIMA DC-5000 treadmill, participants will follow an exercise protocol based on the guidelines of the American College of Sports Medicine (ACSM), consisting of: a 10-minute warm-up, a 20-30-minute loading phase at 40-60% of heart rate reserve (moderate-to-vigorous intensity), and a 10-minute cool-down, all performed at 0% incline.
  Throughout the sessions, participants' heart rate and oxygen saturation levels will be monitored via a fingertip pulse oximeter. Fatigue and dyspnea levels will also be assessed and recorded using the Modified Borg Scale.
  Arms: Traditional Aerobic Exercise Training Group
Other: Aerobic exercise with music therapy — Music Therapy-Based Aerobic Exercise Training group will follow the same treadmill exercise program as the Traditional Aerobic Exercise group. However, during the exercise sessions, music therapy will be applied according to the beats per minute (BPM) ranges specified below: Warm-up (10 minutes, BPM: 80-100): Low-intensity walking accompanied by slow-tempo music Loading Phase (20-30 minutes, BPM: 120-140): Moderate-to-high intensity walking accompanied by rhythmic, motivational music Cool-down (10 minutes, BPM: 80-100): Low-intensity walking accompanied by slow-tempo sedative music Music will be used throughout the exercise sessions to regulate participants' heart rate and blood pressure, reduce perceived fatigue, enhance motivation, and support rhythmic movement patterns. During training, participants' heart rate and oxygen saturation will be monitored using a fingertip pulse oximeter.
  Arms: Music Therapy-Based Aerobic Exercise Training Group

SUMMARY:
The aim of this study is to comparatively evaluate the effects of a music therapy-based aerobic exercise program and traditional aerobic exercise training on cardiopulmonary functions, functional capacity, balance, peripheral muscle strength, cognitive functions, depression level and quality of life in geriatric individuals.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older
* Willingness to participate in the study

Exclusion Criteria:

* Presence of uncontrolled hypertension (≥180/110 mmHg) or severe complications of diabetes (e.g., diabetic neuropathy, proliferative retinopathy, uncontrolled hypoglycemic episodes)
* Presence of respiratory diseases such as Chronic Obstructive Pulmonary Disease (COPD), asthma, etc.
* Presence of chronic neurological disorders such as Multiple Sclerosis (MS), Parkinson's Disease, Amyotrophic Lateral Sclerosis (ALS), etc.
* Diagnosis of any oncological disease
* Presence of acute musculoskeletal conditions that would prevent participation in exercise (e.g., fracture, advanced osteoarthritis, severe musculoskeletal injuries)
* Having undergone any surgical operation within the past 6 months
* Presence of visual or auditory impairments that could interfere with the assessment procedures
* A score of ≤24 on the Mini-Mental State Examination (MMSE), indicating cognitive impairment
* Participation in a regular exercise program within the last six months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate (beats per minute) | 2 months
  There will be important measures to evaluate cardiovascular fitness and exercise responses of geriatric individuals. Heart rate will be dynamically monitored during exercise and will be used to evaluate exercise intensity and cardiovascular responses.
Heart Rate Recovery (beats per minute) | 2 months
  There will be important measures to evaluate cardiovascular fitness and exercise responses of geriatric individuals. Heart rate recovery will be important as an indicator of cardiovascular health by determining the rate at which heart rate returns to normal after exercise and will be measured at 5 and 10 minutes after exercise.
Blood Pressure (mmHg) | 2 months
  Systolic and diastolic blood pressures will be measured using a standard sphygmomanometer to evaluate cardiovascular response to exercise.
Modified Borg Scale Score | 2 months
  Subjective symptoms such as fatigue and dyspnea will be assessed using the Modified Borg Scale during exercise (6-20).
Forced Expiratory Volume in 1 Second (FEV1) (% predicted) | 3 months
  FEV1 refers to the volume of air forcibly exhaled in the first second of a forced breath. It will be measured to evaluate airway obstruction and respiratory capacity, and recorded as a percentage of predicted values based on age, sex, height, and weight. The assessment will be conducted in accordance with American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines using a COSMED MicroQuark spirometer (COSMED, Italy).
Forced Vital Capacity (FVC) (% predicted) | 3 months
  FVC represents the total amount of air exhaled during the spirometry test. It will be used to assess lung volume and capacity, and values will be recorded as a percentage of the predicted normal based on demographic data. Measurements will be performed in compliance with ATS/ERS standards using the COSMED MicroQuark spirometer (COSMED, Italy).
FEV1/FVC Ratio | 3 months
  The FEV1/FVC ratio is a key marker in distinguishing obstructive from restrictive pulmonary patterns. This ratio will be calculated and expressed as a unitless value. Testing will follow ATS/ERS spirometry criteria and be performed using a COSMED MicroQuark spirometer (COSMED, Italy).
Peak Expiratory Flow (PEF) (% predicted) | 3 months
  PEF is the maximum speed of expiration and indicates large airway function. It will be recorded as a percentage of the predicted value and used to monitor bronchial flow capacity and effort. Evaluation will be conducted according to ATS/ERS standards using the COSMED MicroQuark spirometry device (COSMED, Italy).
Forced Expiratory Flow 25-75% (FEF25-75%) (% predicted) | 3 months
  FEF25-75% measures the average flow rate during the middle half of the forced expiration. It reflects small airway function and early signs of airflow limitation, reported as a percentage of predicted normal values. All measurements will be obtained in line with ATS/ERS guidelines using the COSMED MicroQuark spirometer (COSMED, Italy).
Maximum Inspiratory Pressure (MIP) (cmH₂O) | 3 months
  MIP will be measured to evaluate inspiratory muscle strength using a portable electronic intraoral pressure measuring device (MicroRPM, Micro Medical; England), in accordance with ATS and ERS criteria. Participants will perform a maximal inspiratory effort (Müller maneuver) for a few seconds through the mouthpiece, and the highest value will be recorded in cmH₂O.
Maximum Expiratory Pressure (MEP) (cmH₂O) | 3 months
  MEP will be assessed to determine expiratory muscle strength using the same MicroRPM device (Micro Medical; England), following ATS and ERS standards. Participants will perform a maximal expiratory effort (Valsalva maneuver) for a few seconds, and the peak pressure value will be recorded in cmH₂O.
Functional Capacity | 3 months
  The 6-Minute Walk Test (6 DYT) will be used to assess the submaximal functional capacity of the participants. The aim of the 6-Minute Walk Test is to walk the longest distance possible in a 30-meter corridor in 6 minutes. The 6 DYT will be performed in accordance with the guidelines reported by the American Thoracic Society.

SECONDARY OUTCOMES:
Body Weight (kg) | 3 months
  Body weight will be measured using the OMRON BF511 Body Composition Monitor (OMRON Healthcare Co., Japan). Measurements will be taken with participants standing barefoot, wearing light clothing, and the values will be recorded in kilograms.
Height (cm) | 3 months
  Height will be measured with participants standing barefoot, feet together, heels, hips, and head touching the wall, in accordance with standard anthropometric procedures. The value will be entered into the OMRON BF511 Body Composition Monitor for BMI calculation.
Body Mass Index (BMI) (kg/m²) | 3 months
  BMI will be automatically calculated by the OMRON BF511 Body Composition Monitor (OMRON Healthcare Co., Japan) using the entered height and measured weight. It will serve as an indicator of general body composition and nutritional status.
Body Fat Percentage (%) | 3 months
  Body fat percentage will be assessed using the OMRON BF511 Body Composition Monitor (OMRON Healthcare Co., Japan). This parameter will provide insight into total fat mass relative to body weight, contributing to the overall evaluation of body composition.
Skeletal Muscle Ratio (%) | 3 months
  Skeletal muscle ratio will be determined with the OMRON BF511 Body Composition Monitor (OMRON Healthcare Co., Japan). It will represent the percentage of skeletal muscle mass in relation to total body mass and be used to assess muscular health and function.
Basal Metabolic Rate (BMR) (kcal/day) | 3 months
  Basal Metabolic Rate will be measured in kilocalories per day using the OMRON BF511 Body Composition Monitor (OMRON Healthcare Co., Japan). This value reflects the daily energy expenditure at rest and will be used to assess metabolic function.
Postural Stability | 3 months
  Postural stability will be assessed using the "Postural Stability Test" module of the Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA). This test evaluates the ability to maintain a stable position on a static or dynamic platform. Higher scores indicate poorer balance performance, and results will be used to assess static and dynamic postural control.
Limits of Stability | 3 months
  The "Limits of Stability Test" on the Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA) will measure the participant's ability to voluntarily shift their center of gravity toward various directions without losing balance. A lower score represents better dynamic balance and postural control.
Clinical Test of Sensory Integration of Balance | 3 months
  The "Clinical Test of Sensory Integration of Balance" will be performed using the Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA) to evaluate how the somatosensory, visual, and vestibular systems contribute to postural stability. This score helps determine the sensory system impairments affecting balance, with higher scores reflecting greater postural sway and reduced sensory integration.
Handgrip Strength | 3 months
  Handgrip strength will be assessed for upper extremity muscle strength assessment. This assessment will be performed on the dominant hand with a hydraulic hand dynamometer (JAMAR hydraulic hand dynamometer, ABD) and each measurement will be repeated 3 times to determine the maximum grip strength and the average will be recorded.
Timed Up and Go Test (TUG) | 3 months
  Lower extremity muscle strength and fall risk assessment will be performed with the "Timed Up and Go Test (TUG)". Participants will be asked to get up from a chair with a seat height of approximately 46 cm, walk 3 meters and sit down again, the completed time will be recorded in seconds.
30 Second Sit-to-Stand Test | 3 months
  The "30 Second Sit-to-Stand Test" will be used for lower extremity muscle strength assessment. Participants will be asked to get up and sit down from a chair with their hands crossed on their chest for 30 seconds with as many repetitions as possible.
Physical Activity | 3 months
  Physical activity level will be assessed with the "Physical Activity Scale for the Elderly (PASE)". "PASE" assesses the physical activity of elderly individuals in the last week. Participation in leisure time activities, housework and work-related activities is recorded in the scale. There are options for the duration of the activity as less than 1 hour, between 1 and 2 hours, 2-4 hours or more than 4 hours. Paid or unpaid work-related activities are recorded as total hours per week. Housework activities (light and heavy); gardening, home repairs, outdoor activities and activities related to caring for others are expressed with the options 'Yes' and 'No'. The calculation of the total score of the scale is carried out by multiplying the time spent on each activity (hours/week) or participation in an activity (yes/no) by the item values and summing the scores of all activities.
Depression | 3 months
  Depression assessment will be performed with the "Geriatric Depression Scale-15 (GDS-15)". The "Geriatric Depression Scale-15" is a depression scale developed for the elderly population. It is prepared in a way that elderly individuals can answer "yes" or "no", consisting of a total of 15 questions. In the evaluation of the scale, 1 point is given for each yes answer in favor of depression, and 0 points are given for a no answer. The total score obtained from the scale is accepted as the depression score. The scale is scored as follows; 0-10 points as "no depression", 11-13 points as "possible depression", and 14 and above as "definite depression". When the threshold value for the "Geriatric Depression Scale-15" scores is taken as 14, its specificity approaches 100%.
Quality of Life Assessment | 3 months
  Quality of life will be assessed with the "Quality of Life Scale in the Elderly - Short Form". This scale was developed by Bowling and his colleagues to be used in the assessment of quality of life in the geriatric population. In the single item asked at the beginning of the test, the person is asked to score their quality of life as 1-very bad and 5-very good, but this score is not evaluated together with the total scale score. For each item, answers are given as 1-strongly disagree and 5-strongly agree and consist of a total of 13 items. The total score is calculated between 13-65. Higher scores indicate better quality of life.
Cognitive Functions | 3 months
  The Montreal Cognitive Assessment Scale (MoCA) will be used to evaluate cognitive functions. MoCA is a questionnaire developed to evaluate different cognitive functions and mild cognitive impairment. The cognitive functions evaluated in the test are; memory, concentration, memory, language, abstract thinking, orientation, calculation, visual structuring and executive functions. The maximum score that the patient can obtain from the test is 30, a score of 21 or above will be considered as no mild cognitive impairment.
Exercise Enjoyment | 3 months
  Participants' enjoyment of exercise will be assessed with the "Exercise Enjoyment Scale". Each item is assessed on a scale of 1 to 7 points, with a neutral point of four indicating how much the participant enjoys the exercise, based on the participant's response to the question "How do you feel about the exercise you are currently doing?" The higher the score the participant will receive from the scale, the more they enjoy the physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Can Törpü, PhD(c), Principal Investigator — Bezmialem Vakif University; Alis Kostanoğlu, PhD, Study Director — Bezmialem Vakif University; Muhammed Tunç, MD, Study Chair — Bezmialem Vakif University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park KS, Buseth L, Hong J, Etnier JL. Music-based multicomponent exercise training for community-dwelling older adults with mild-to-moderate cognitive decline: a feasibility study. Front Med (Lausanne). 2023 Aug 21;10:1224728. doi: 10.3389/fmed.2023.1224728. eCollection 2023. PMID 37671396
- [Background] Chan SY, Chen CF. Effects of an Active Music Therapy Program on Functional Fitness in Community Older Adults. J Nurs Res. 2020 Oct;28(5):e111. doi: 10.1097/JNR.0000000000000391. PMID 32649395
- [Background] Trombetti A, Hars M, Herrmann FR, Kressig RW, Ferrari S, Rizzoli R. Effect of music-based multitask training on gait, balance, and fall risk in elderly people: a randomized controlled trial. Arch Intern Med. 2011 Mar 28;171(6):525-33. doi: 10.1001/archinternmed.2010.446. Epub 2010 Nov 22. PMID 21098340
- [Background] Estebsari F, Dastoorpoor M, Khalifehkandi ZR, Nouri A, Mostafaei D, Hosseini M, Esmaeili R, Aghababaeian H. The Concept of Successful Aging: A Review Article. Curr Aging Sci. 2020;13(1):4-10. doi: 10.2174/1874609812666191023130117. PMID 31657693